CLINICAL TRIAL: NCT05222659
Title: Perioperative Glucose and Insulin Changes in Major Urologic Surgeries
Acronym: PEGLINS
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Jill Hamilton-Reeves, PhD RD LD, Associate Professor, University of Kansas Medical Center
Other Study IDs: STUDY00147628
Record Dates: First submitted 2022-01-13; First posted 2022-02-03 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Urologic Diseases; Surgery; Blood Glucose, High
Keywords: surgery, blood glucose, continuous glucose monitoring
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Urologic surgery patients

SUMMARY:
Urological surgery patients will have their blood glucose measured before, during, and after surgery. Blood glucose will be measured using a continuous glucose monitor (CGM) device. We hypothesize the presence of a hyperglycemic state towards the end of surgery due to increased metabolic demand.

DETAILED DESCRIPTION:
Surgical stress causes acute insulin resistance, increased circulating free-fatty acids, and reduced blood glucose uptake resulting in hyperglycemia. Intraoperative and postoperative glucose levels are typically only monitored in the diabetic or cardiac surgical patient. There is a lack of data on perioperative glucose levels in most prolonged surgeries and thus a barrier in determining the best glycemic management strategy to prevent or resolve acute insulin resistance and hyperglycemia. Obtaining blood glucose by CGM is less invasive and will avert disruption of current surgical pathways and standards of care while also producing reliable glucose measurements.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years) undergoing a major urologic surgery (proposed case duration >4 hours) at The University of Kansas Medical Center (KUMC)
* English speaking

Exclusion Criteria:

* Diagnosis of Type 1 or Type 2 diabetes mellitus or an A1C > 6.5%
* Pregnant or lactating
* Known allergy to milk, soy, egg, wheat, peanuts, or tree nuts
* Swallowing difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing major urologic surgery at KUMC
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
To determine the perioperative glycemic changes longitudinally in patients undergoing major urologic surgeries. | Perioperatively up to post-operative day 4
  Interstitial blood glucose levels measured by Continuous Glucose Monitor (CGM) device, in mg/dL

SECONDARY OUTCOMES:
To determine the effect of perioperative insulin levels on glycemic variations in patients undergoing major urologic surgeries. | Perioperatively up to post-operative day 4
  Serum insulin in uIU/mL will be measured from participant blood samples
To determine the effect of perioperative insulin, C-peptide, and Free-Fatty Acid (FFA) | Perioperatively up to post-operative day 4
  C-peptide in ng/mL will be measured from participant blood samples
To determine the effect of perioperative insulin, C-peptide, and Free-Fatty Acid (FFA) | Perioperatively up to post-operative day 4
  FFA in mmol/L will be measured from participant blood samples

OTHER OUTCOMES:
To determine gastric emptying time of a carbohydrate drink. | at least 2 days before surgery
  A specialized carbohydrate beverage will be given to a subset of willing participants in order to establish a feasible interval for consumption before surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jill Hamilton-Reeves, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No